CLINICAL TRIAL: NCT01308034
Title: Phase I Study of Continuous Dosing of Sunitinib in Non GIST Sarcomas With Concomitant Radiotherapy
Brief Title: Study of Continuous Dosing of Sunitinib in Non GIST Sarcomas With Concomitant Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT - SUTENT; 2010-021551-11 (EudraCT Number)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Non GIST Sarcomas
Keywords: non GIST sarcomas; sunitinib; radiotherapy; dose escalation
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- association sunitinib radiotherapy (Experimental)
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — All patients will be treated with sunitinib (2 dose levels) once a day (in the morning) for 6 weeks in association with radiotherapy.Radiotherapy will be realised 1-4h after taking sunitinib.
  Dose level 1 : 25 mg once daily Dose level 2 : 37.5 mg once daily Authorization to include a patient in the upper step will be given only if the deadline of 14 weeks after the start of treatment of last patient included were strictly respected and depending of number of DLT occuring.

SUMMARY:
The purpose of this study is to determine the safety of continuous dosing of sunitinib in association with radiotherapy in patients with non GIST (gastro intestinal stromal tumor) sarcomas who cannot be treated by surgery.

The primary objective of the study is to determine the maximum tolerated dose (MTD) of continuous dosing of sunitinib in association with radiotherapy in patients with non GIST sarcomas who cannot be treated by surgery.

This study is a multicentre, open-label phase I with dose escalation : 2 dose levels.

3-6 patients will be included at each dose level.3-18 patients will be included in the study.

DETAILED DESCRIPTION:
Study design : 2 dose levels

Step 1 : 25 mg once daily Step 2 : 37.5 mg once daily

3-6 patients will be included at each of the sunitinib dose levels, depending on the number of DLTs (dose limiting toxicity) occurring in 14 weeks after start of treatment

DLT is defined as :

any grade 3 or 4 musculoskeletal or cutaneous toxicity within the field of radiation any other toxicity > or = 4

Secondary objectives are :

* to evaluate the safety with late toxicities
* to estimate the response rate at 6 months
* to estimate the progression free survival
* to evaluate the proportion of patients with an operable tumour after treatment

Exploratory objectives are :

* to study evolution during treatment of neo-angiogenesis measured by dynamic contrast enhanced-ultrasonography (DCE-US)
* to study the correlation between clinical response and changes of tumor perfusion measured by DCE-US

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years of age
2. Histologically or cytologically (in case of recurrence) confirmed connective tissue neoplasm, including any of the following subtypes:

   * Liposarcomas
   * Fibrosarcoma, myxofibrosarcoma
   * Undifferentiated pleomorphic sarcoma
   * Leiomyosarcomas
   * Pleomorphic rhabdomyosarcomas only
   * Angiosarcomas
   * Uncertain differentiated tumors: synovial sarcomas, epithelioid sarcomas, alveolar sarcomas, clear cells sarcomas.

   or osteosarcoma diagnosis, chondrosarcoma or chordoma.
3. Locally advanced or locally recurrent inoperable tumor without previous irradiation [inoperable status must be assessed by staff including a surgeon specialized in sarcoma].
4. No prior treatment by sunitinib malate
5. Life expectancy > 6 months
6. ECOG performance status ≤ 2
7. Blood tests, renal and liver functions in the normal range with, in the 7 days prior to study entry, blood or serum values as follows:

   * Absolute neutrophil count ≥ 1.,5 G/L
   * Platelet count ≥ 100 G/L
   * Bilirubin ≤ 1.5 mg/dL
   * PT and INR ≤ 1.5 times upper limit of normal [Patients under preventive anticoagulant therapy are allowed to participate]
   * AST and ALT ≤ 2.5 times upper limit of normal
   * Creatinine ≤ 150 umol/L
   * Calcium ≤ 12 mg/dL
   * Blood glucose < 150 mg/dL
8. Fertile patients must use effective contraception prior to, during, and for 28 days after completion of study therapy
9. Ability to swallow oral medications
10. Mandatory affiliation with a health insurance company
11. Signed written informed consent.

Exclusion Criteria:

1. GIST, Ewing sarcoma or embryonic rhabdomyosarcomas
2. Radiation field including lung, bowel, or central nervous system
3. Pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication
4. NCI grade ≥ 3 hemorrhage within the past 4 weeks prior to study drug administration
5. Significant cardiovascular disease (New York Heart Association (NYHA) > grade 2 congestive cardiac failure, myocardial infarction within 6 months prior to inclusion, unstable angina, severe cardiac arrhythmia, severe cerebrovascular accident within 6 months prior to inclusion, history of severe thromboembolism (pulmonary embolism or deep vein thrombosis DVT) within 6 months prior to inclusion (patients with recent history of DVT treated by anticoagulant (except therapeutic warfarin)during at least 6 weeks are eligibles), prolonged QTc interval (QTc > 480 msec with Bazett), bradycardia (heart rate < 45bpm), electrolytic troubles (hyponatremia<120mmol/l, kalemia≥6mmol/l) or uncontrolled hypertension while receiving appropriate medication (≥ 160 mm Hg systolic and/or ≥ 90 mm Hg diastolic).
6. Less than 6 weeks between prior neoplastic treatment by tyrosine kinase inhibitor and inclusion and less than 4 weeks for other neoplastic treatments
7. Major surgical procedure, open biopsy, or serious non healing wound within 28 days prior to first day of treatment
8. Concurrent participation in another clinical trial
9. Other disease or illness within the past 6 months prior to study drug administration, including the following:

   * Psychiatric illness or social situation that would preclude study compliance
   * Known human immunodeficiency virus (HIV)- or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
10. Known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease
11. peritoneal carcinosis
12. number of metastatic sites > 2
13. Restriction of freedom by judicial or administrative decision
14. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2016-05 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
the number of DLT occurring at each dose level of sunitinib within 14 weeks after the start of treatment | within 14 weeks after the start of treatment

SECONDARY OUTCOMES:
the number of early toxicities (within 14 weeks after the beginning of treatment) and late toxicities (after 14 weeks and until 12 months after the start of treatment) using NCI-CTC v3.0 and RTOG-EORTC | within 12 months after the start of treatment
response rate at 6 months using MRI (magnetic resonance imaging) | 6 months after the start of treatment
progression free survival measured from the date of inclusion to the date of first evidence of progression or date of death of any cause, or to the date of last follow up | within 12 months after the start of treatment
evolution of neo-angiogenesis during treatment measured by DCE-US | within 6 weeks after the start of treatment
correlation between clinical response and change of tumor perfusion measured by DCE-US | within 12 months after the start of treatment
proportion of patients operable after treatment | at week 6 after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Blay, PR, Principal Investigator — Centre Léon Bérard, Lyon; Marie Pierre Sunyach, Principal Investigator — Centre Léon Bérard, Lyon
Locations (6):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - Institut de Cancérologie de l'ouest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Alektiar KM, Velasco J, Zelefsky MJ, Woodruff JM, Lewis JJ, Brennan MF. Adjuvant radiotherapy for margin-positive high-grade soft tissue sarcoma of the extremity. Int J Radiat Oncol Biol Phys. 2000 Nov 1;48(4):1051-8. doi: 10.1016/s0360-3016(00)00753-7. PMID 11072162
- [Background] Zagars GK, Ballo MT. Significance of dose in postoperative radiotherapy for soft tissue sarcoma. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):473-81. doi: 10.1016/s0360-3016(02)04573-x. PMID 12738323
- [Background] Tepper JE, Suit HD. Radiation therapy alone for sarcoma of soft tissue. Cancer. 1985 Aug 1;56(3):475-9. doi: 10.1002/1097-0142(19850801)56:33.0.co;2-s. PMID 4005809
- [Background] Schwartz DL, Einck J, Bellon J, Laramore GE. Fast neutron radiotherapy for soft tissue and cartilaginous sarcomas at high risk for local recurrence. Int J Radiat Oncol Biol Phys. 2001 Jun 1;50(2):449-56. doi: 10.1016/s0360-3016(00)01586-8. PMID 11380233
- [Background] Schmitt G, Pape H, Zamboglou N. Long term results of neutron- and neutron-boost irradiation of soft tissue sarcomas. Strahlenther Onkol. 1990 Jan;166(1):61-2. PMID 2154050
- [Background] Alektiar KM, Brennan MF, Healey JH, Singer S. Impact of intensity-modulated radiation therapy on local control in primary soft-tissue sarcoma of the extremity. J Clin Oncol. 2008 Jul 10;26(20):3440-4. doi: 10.1200/JCO.2008.16.6249. PMID 18612160
- [Background] Donnay L, Dejean C, Amsellem E, Bourezgui H, de Figueiredo BH, Duparc A, Caron J, Tournat H, Lagarde P, Stoeckle E, Kantor G. [Radiotherapy for soft tissue sarcomas of extremities. Preliminary comparative dosimetric study of 3D conformal radiotherapy versus helical tomotherapy]. Cancer Radiother. 2008 Dec;12(8):809-16. doi: 10.1016/j.canrad.2008.08.275. Epub 2008 Nov 28. French. PMID 19046919
- [Background] Folkman J. The role of angiogenesis in tumor growth. Semin Cancer Biol. 1992 Apr;3(2):65-71. PMID 1378311
- [Background] Jain RK. Normalization of tumor vasculature: an emerging concept in antiangiogenic therapy. Science. 2005 Jan 7;307(5706):58-62. doi: 10.1126/science.1104819. PMID 15637262
- [Background] Overgaard J, Horsman MR. Modification of Hypoxia-Induced Radioresistance in Tumors by the Use of Oxygen and Sensitizers. Semin Radiat Oncol. 1996 Jan;6(1):10-21. doi: 10.1053/SRAO0060010. PMID 10717158
- [Background] Overgaard J. Hypoxic radiosensitization: adored and ignored. J Clin Oncol. 2007 Sep 10;25(26):4066-74. doi: 10.1200/JCO.2007.12.7878. PMID 17827455
- [Background] Hess C, Vuong V, Hegyi I, Riesterer O, Wood J, Fabbro D, Glanzmann C, Bodis S, Pruschy M. Effect of VEGF receptor inhibitor PTK787/ZK222584 [correction of ZK222548] combined with ionizing radiation on endothelial cells and tumour growth. Br J Cancer. 2001 Dec 14;85(12):2010-6. doi: 10.1054/bjoc.2001.2166. PMID 11747347
- [Background] Lee CG, Heijn M, di Tomaso E, Griffon-Etienne G, Ancukiewicz M, Koike C, Park KR, Ferrara N, Jain RK, Suit HD, Boucher Y. Anti-Vascular endothelial growth factor treatment augments tumor radiation response under normoxic or hypoxic conditions. Cancer Res. 2000 Oct 1;60(19):5565-70. PMID 11034104
- [Background] Li J, Huang S, Armstrong EA, Fowler JF, Harari PM. Angiogenesis and radiation response modulation after vascular endothelial growth factor receptor-2 (VEGFR2) blockade. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1477-85. doi: 10.1016/j.ijrobp.2005.04.028. PMID 16029810
- [Background] Cao C, Albert JM, Geng L, Ivy PS, Sandler A, Johnson DH, Lu B. Vascular endothelial growth factor tyrosine kinase inhibitor AZD2171 and fractionated radiotherapy in mouse models of lung cancer. Cancer Res. 2006 Dec 1;66(23):11409-15. doi: 10.1158/0008-5472.CAN-06-2414. PMID 17145887
- [Background] Dings RP, Loren M, Heun H, McNiel E, Griffioen AW, Mayo KH, Griffin RJ. Scheduling of radiation with angiogenesis inhibitors anginex and Avastin improves therapeutic outcome via vessel normalization. Clin Cancer Res. 2007 Jun 1;13(11):3395-402. doi: 10.1158/1078-0432.CCR-06-2441. PMID 17545548
- [Background] Riesterer O, Honer M, Jochum W, Oehler C, Ametamey S, Pruschy M. Ionizing radiation antagonizes tumor hypoxia induced by antiangiogenic treatment. Clin Cancer Res. 2006 Jun 1;12(11 Pt 1):3518-24. doi: 10.1158/1078-0432.CCR-05-2816. PMID 16740778
- [Background] Williams KJ, Telfer BA, Brave S, Kendrew J, Whittaker L, Stratford IJ, Wedge SR. ZD6474, a potent inhibitor of vascular endothelial growth factor signaling, combined with radiotherapy: schedule-dependent enhancement of antitumor activity. Clin Cancer Res. 2004 Dec 15;10(24):8587-93. doi: 10.1158/1078-0432.CCR-04-1147. PMID 15623642
- [Background] Winkler F, Kozin SV, Tong RT, Chae SS, Booth MF, Garkavtsev I, Xu L, Hicklin DJ, Fukumura D, di Tomaso E, Munn LL, Jain RK. Kinetics of vascular normalization by VEGFR2 blockade governs brain tumor response to radiation: role of oxygenation, angiopoietin-1, and matrix metalloproteinases. Cancer Cell. 2004 Dec;6(6):553-63. doi: 10.1016/j.ccr.2004.10.011. PMID 15607960
- [Background] Gaffney DK, Haslam D, Tsodikov A, Hammond E, Seaman J, Holden J, Lee RJ, Zempolich K, Dodson M. Epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF) negatively affect overall survival in carcinoma of the cervix treated with radiotherapy. Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):922-8. doi: 10.1016/s0360-3016(03)00209-8. PMID 12829126
- [Background] Gorski DH, Beckett MA, Jaskowiak NT, Calvin DP, Mauceri HJ, Salloum RM, Seetharam S, Koons A, Hari DM, Kufe DW, Weichselbaum RR. Blockage of the vascular endothelial growth factor stress response increases the antitumor effects of ionizing radiation. Cancer Res. 1999 Jul 15;59(14):3374-8. PMID 10416597
- [Background] Kermani P, Leclerc G, Martel R, Fareh J. Effect of ionizing radiation on thymidine uptake, differentiation, and VEGFR2 receptor expression in endothelial cells: the role of VEGF(165). Int J Radiat Oncol Biol Phys. 2001 May 1;50(1):213-20. doi: 10.1016/s0360-3016(01)01445-6. PMID 11316566
- [Background] Garcia-Barros M, Paris F, Cordon-Cardo C, Lyden D, Rafii S, Haimovitz-Friedman A, Fuks Z, Kolesnick R. Tumor response to radiotherapy regulated by endothelial cell apoptosis. Science. 2003 May 16;300(5622):1155-9. doi: 10.1126/science.1082504. PMID 12750523
- [Background] Gloe T, Sohn HY, Meininger GA, Pohl U. Shear stress-induced release of basic fibroblast growth factor from endothelial cells is mediated by matrix interaction via integrin alpha(v)beta3. J Biol Chem. 2002 Jun 28;277(26):23453-8. doi: 10.1074/jbc.M203889200. Epub 2002 Apr 25. PMID 11976347
- [Background] Bao S, Wu Q, McLendon RE, Hao Y, Shi Q, Hjelmeland AB, Dewhirst MW, Bigner DD, Rich JN. Glioma stem cells promote radioresistance by preferential activation of the DNA damage response. Nature. 2006 Dec 7;444(7120):756-60. doi: 10.1038/nature05236. Epub 2006 Oct 18. PMID 17051156
- [Background] Maki RG, D'Adamo DR, Keohan ML, Saulle M, Schuetze SM, Undevia SD, Livingston MB, Cooney MM, Hensley ML, Mita MM, Takimoto CH, Kraft AS, Elias AD, Brockstein B, Blachere NE, Edgar MA, Schwartz LH, Qin LX, Antonescu CR, Schwartz GK. Phase II study of sorafenib in patients with metastatic or recurrent sarcomas. J Clin Oncol. 2009 Jul 1;27(19):3133-40. doi: 10.1200/JCO.2008.20.4495. Epub 2009 May 18. PMID 19451436
- [Background] Basso U, Brunello A, Bertuzzi A, Santoro A. Sorafenib is active on lung metastases from synovial sarcoma. Ann Oncol. 2009 Feb;20(2):386-7. doi: 10.1093/annonc/mdn685. No abstract available. PMID 19211500
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] George S, Merriam P, Maki RG, Van den Abbeele AD, Yap JT, Akhurst T, Harmon DC, Bhuchar G, O'Mara MM, D'Adamo DR, Morgan J, Schwartz GK, Wagner AJ, Butrynski JE, Demetri GD, Keohan ML. Multicenter phase II trial of sunitinib in the treatment of nongastrointestinal stromal tumor sarcomas. J Clin Oncol. 2009 Jul 1;27(19):3154-60. doi: 10.1200/JCO.2008.20.9890. Epub 2009 May 18. PMID 19451429
- [Background] Crane CH, Eng C, Feig BW, Das P, Skibber JM, Chang GJ, Wolff RA, Krishnan S, Hamilton S, Janjan NA, Maru DM, Ellis LM, Rodriguez-Bigas MA. Phase II trial of neoadjuvant bevacizumab, capecitabine, and radiotherapy for locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):824-30. doi: 10.1016/j.ijrobp.2009.02.037. Epub 2009 May 21. PMID 19464823
- [Background] Koukourakis MI, Giatromanolaki A, Sheldon H, Buffa FM, Kouklakis G, Ragoussis I, Sivridis E, Harris AL; Tumour and Angiogenesis Research Group. Phase I/II trial of bevacizumab and radiotherapy for locally advanced inoperable colorectal cancer: vasculature-independent radiosensitizing effect of bevacizumab. Clin Cancer Res. 2009 Nov 15;15(22):7069-76. doi: 10.1158/1078-0432.CCR-09-0688. Epub 2009 Nov 3. PMID 19887481
- [Background] Lordick F, Geinitz H, Theisen J, Sendler A, Sarbia M. Increased risk of ischemic bowel complications during treatment with bevacizumab after pelvic irradiation: report of three cases. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1295-8. doi: 10.1016/j.ijrobp.2005.12.004. Epub 2006 Feb 28. PMID 16503384
- [Background] Crane CH, Winter K, Regine WF, Safran H, Rich TA, Curran W, Wolff RA, Willett CG. Phase II study of bevacizumab with concurrent capecitabine and radiation followed by maintenance gemcitabine and bevacizumab for locally advanced pancreatic cancer: Radiation Therapy Oncology Group RTOG 0411. J Clin Oncol. 2009 Sep 1;27(25):4096-102. doi: 10.1200/JCO.2009.21.8529. Epub 2009 Jul 27. PMID 19636002
- [Background] Lai A, Filka E, McGibbon B, Nghiemphu PL, Graham C, Yong WH, Mischel P, Liau LM, Bergsneider M, Pope W, Selch M, Cloughesy T. Phase II pilot study of bevacizumab in combination with temozolomide and regional radiation therapy for up-front treatment of patients with newly diagnosed glioblastoma multiforme: interim analysis of safety and tolerability. Int J Radiat Oncol Biol Phys. 2008 Aug 1;71(5):1372-80. doi: 10.1016/j.ijrobp.2007.11.068. Epub 2008 Mar 20. PMID 18355978
- [Background] Gutin PH, Iwamoto FM, Beal K, Mohile NA, Karimi S, Hou BL, Lymberis S, Yamada Y, Chang J, Abrey LE. Safety and efficacy of bevacizumab with hypofractionated stereotactic irradiation for recurrent malignant gliomas. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):156-63. doi: 10.1016/j.ijrobp.2008.10.043. Epub 2009 Jan 23. PMID 19167838
- [Background] Schueneman AJ, Himmelfarb E, Geng L, Tan J, Donnelly E, Mendel D, McMahon G, Hallahan DE. SU11248 maintenance therapy prevents tumor regrowth after fractionated irradiation of murine tumor models. Cancer Res. 2003 Jul 15;63(14):4009-16. PMID 12873999
- [Background] Cuneo KC, Geng L, Fu A, Orton D, Hallahan DE, Chakravarthy AB. SU11248 (sunitinib) sensitizes pancreatic cancer to the cytotoxic effects of ionizing radiation. Int J Radiat Oncol Biol Phys. 2008 Jul 1;71(3):873-9. doi: 10.1016/j.ijrobp.2008.02.062. PMID 18514780
- [Background] Kao J, Packer S, Vu HL, Schwartz ME, Sung MW, Stock RG, Lo YC, Huang D, Chen SH, Cesaretti JA. Phase 1 study of concurrent sunitinib and image-guided radiotherapy followed by maintenance sunitinib for patients with oligometastases: acute toxicity and preliminary response. Cancer. 2009 Aug 1;115(15):3571-80. doi: 10.1002/cncr.24412. PMID 19536893
- [Result] Rosenberg SA, Tepper J, Glatstein E, Costa J, Baker A, Brennan M, DeMoss EV, Seipp C, Sindelar WF, Sugarbaker P, Wesley R. The treatment of soft-tissue sarcomas of the extremities: prospective randomized evaluations of (1) limb-sparing surgery plus radiation therapy compared with amputation and (2) the role of adjuvant chemotherapy. Ann Surg. 1982 Sep;196(3):305-15. doi: 10.1097/00000658-198209000-00009. PMID 7114936
- [Result] Harrison LB, Franzese F, Gaynor JJ, Brennan MF. Long-term results of a prospective randomized trial of adjuvant brachytherapy in the management of completely resected soft tissue sarcomas of the extremity and superficial trunk. Int J Radiat Oncol Biol Phys. 1993 Sep 30;27(2):259-65. doi: 10.1016/0360-3016(93)90236-o. PMID 8407399
- [Result] Yang JC, Chang AE, Baker AR, Sindelar WF, Danforth DN, Topalian SL, DeLaney T, Glatstein E, Steinberg SM, Merino MJ, Rosenberg SA. Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol. 1998 Jan;16(1):197-203. doi: 10.1200/JCO.1998.16.1.197. PMID 9440743